CLINICAL TRIAL: NCT04319874
Title: Phase II Clinical Trial Scheme of Ganoderma Lucidum Spore Powder for Postoperative Chemotherapy of Osteosarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YANWQ003
Record Dates: First submitted 2020-03-16; First posted 2020-03-24 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Osteosarcoma
Keywords: Ganoderma lucidum; osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — Drug Therapy; Neoadjuvant Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- sham group (Sham Comparator): Treated with conventional chemotherapy drugs
  Interventions: Drug: Chemotherapy
- NC group (Placebo Comparator): Treated with conventional chemotherapy drugs and Placebo
  Interventions: Drug: Chemotherapy; Drug: Placebos
- experimental group (Experimental): Treated with conventional chemotherapy drugs and Ganoderma lucidum
  Interventions: Drug: Ganoderma lucidum; Drug: Chemotherapy

INTERVENTIONS:
Drug: Ganoderma lucidum — Participants take ganoderma lucidum spore powder once a day, 1000mg
  Other Names: lingzhi trearment
  Arms: experimental group
Drug: Chemotherapy — Subjects are treated with conventional chemotherapy
  Other Names: Chemotherapy treatment
Drug: Placebos — Subjects are treated with conventional chemotherapy and Placebos once a day, 1000mg
  Other Names: PLacebos treatment
  Arms: NC group

SUMMARY:
Osteosarcoma is the most common primary highly malignant bone tumor in children and young people. Incidence rates are bimodal, with the first peak occurring in adolescence and the second peak in patients over 60 years of age. The 5-year survival rate of patients with osteosarcoma is less than 20%. This study aims to improve the prognosis of patients and change the outcome of patients with osteosarcoma.

DETAILED DESCRIPTION:
This project intends to conduct a multicenter, randomized, double-blind, parallel-controlled clinical trial of ganoderma spore powder and doxorubicin combined with cisplatin chemotherapy in the treatment of osteosarcoma patients. The combination therapy of traditional chemotherapeutics has not played a good effect and has large side effects. The Ganoderma lucidum spore powder group is a natural botanical drug that has a good anti-tumor auxiliary effect in regulating the tumor immune microenvironment. The investigators' previous research showed that Ganoderma lucidum spore powder can inhibit the growth and metastasis of osteosarcoma in the body without obvious toxic and side effects, which indicates that this research scheme has strong feasibility.

ELIGIBILITY:
Inclusion Criteria:

- Signed informed consent form

Clinical diagnosis of osteosarcoma

Must be able to swallow tablets

after surgical resection

Exclusion Criteria:

- Symptomatic central nervous system metastases and/or carcinomatous meningitis Known HIV or active hepatitis B/C infection

Active infection requiring systemic treatment

Clinically significant cardiac arrhythmias

Class III or IV Congestive Heart Failure as defined by the New York Heart

Association functional classification system < 6 months prior to screening

A pregnant or nursing female, or women of child-bearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception

Any condition for which participation would not be in the best interest of the participant

Patients unable to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures or those with severe psychiatric illness/social situations that would limit compliance with study requirements

Patients participating in another clinical investigation at the time of signature of the informed consent

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-09-15 (Estimated); Primary Completion 2022-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Effect of 5-year survival rate of Ganoderma osteosarcoma patients | up to 60 months
  Karnofsky (Karlfeld, KPS, percentile) functional status scoring criteria

IPD SHARING:
Plan to Share IPD: No